CLINICAL TRIAL: NCT07281365
Title: Proof-of-Concept Trial of an Emotion Regulation and Executive Functioning Intervention for SITBs in Children
Brief Title: Pilot Trial of an Emotion Regulation and Executive Functioning Intervention for Self-Injurious Thoughts and Behaviors (SITBs) in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-1783; R34MH135963 (NIH)
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Self-injury; Suicidal Ideation and Behavior; Executive Functioning; Emotion Regulation
Keywords: Preadolescents; Children; Self-Injury; Suicidal ideation and behavior; Randomized controlled trial; Feasibility
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Behavior; Emotional Regulation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preadolescent SITB Intervention (Experimental): Experimental intervention for preadolescent SITBs targeting executive functioning, emotion regulation, and other SITB risk factors
  Interventions: Behavioral: Preadolescent SITB Intervention
- Treatment as Usual (TAU) (Active Comparator): Treatment as Usual provided by outpatient mental health therapist
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Treatment as usual (TAU) — Typical interventions Outpatient therapist would provide to a preadolescent with SITBs, based on their clinical judgement
  Arms: Treatment as Usual (TAU)
Behavioral: Preadolescent SITB Intervention — Experimental intervention developed with end-users and experts to target emotion regulation, executive functioning, and other risk factors for SITBs in preadolescents
  Arms: Preadolescent SITB Intervention

SUMMARY:
The goal of this study is to develop and test an outpatient intervention for preadolescents (ages 7-12) with self-injurious thoughts and behaviors (SITBs).

The main questions it aims to answer are:

1. Does the newer intervention lead to better engagement of families in treatment compared to treatment as usual (TAU)?
2. Is the new intervention feasible, acceptable, and appropriate?
3. Does the new intervention lead to more improvements in SITBs, mental health symptoms, and treatment targets compared to TAU?

Preadolescent participants with SITBs and their families will be randomized to either the new intervention or TAU, which will consist of the typical interventions the study therapist would use for preadolescents with SITBs. Participants will:

1. Complete an initial baseline assessment to determine eligibility and assess SITBs, mental health symptoms, executive functioning, and emotion regulation
2. Participate in a ~weekly, outpatient intervention lasting around 3-4 months
3. Complete additional assessments at mid-treatment, post-treatment, and 3-month follow-up
4. Participate in an interview sharing their perceptions of the intervention

DETAILED DESCRIPTION:
In Phase 1 of the study (Aim 1), the investigators will iteratively design an intervention for preadolescent SITBs through a step-by-step process using frameworks for systematically developing and adapting interventions (Wingood et al., 2008; Bartholomew et al., 1998). The design process will incorporate user-centered design methods, whereby multisectoral experts and end-users (i.e., therapists and families) will participate in the design process to maximize the intervention's dissemination and implementation potential. In Phase 2 of the study (Aims 2 and 3), the investigators will conduct a pilot randomized controlled trial (RCT) of the intervention, with a treatment as usual (TAU) comparator, in 52 preadolescents ages 7-12. Aim 2 will evaluate engagement (primary outcome), feasibility, acceptability, and implementation outcomes for the intervention and study procedures. Aim 3 will be to collect preliminary evidence to explore superiority of the SITB intervention to TAU in reducing SITBs and engaging the target mechanisms of EF and emotion regulation.

In Phase 1, the investigators will use mixed methods approaches and user-centered design principles to iteratively develop the preadolescent SITB intervention. Through a needs assessment, the investigators will use an exploratory sequential qualitative--> quantitative mixed methods design, whereby qualitative interviews with therapists will inform the development of a quantitative survey assessing needs and experiences of therapists treating preadolescents with SITBs. Results from the therapist assessment will be integrated with findings from qualitative interviews with preadolescents and caregiversto further inform initial decisions about core functions and specific components of the intervention. During a pre-testing phase utilizing a concurrent mixed methods approach, therapists and preadolescents/families will participate in think-aloud design sessions to provide quantitative and qualitative feedback about rough intervention prototypes. An initial draft of the intervention will then be produced and reviewed by a group of experts, resulting in a second draft of the intervention and therapist training and consultation procedures. A single-arm, pilot feasibility trial of the intervention with 9 preadolescents (ADAPT-ITT Step 8, Part 1) will inform adaptations to the intervention, therapist training, and trial procedures.

Phase 2 will involve training therapists in the intervention, using procedures and materials refined during the pilot trial, followed by a RCT with a TAU control condition with 52 preadolescents (ADAPT-ITT Step 8, Part 2). The trial will be powered to detect differences in engagement between conditions (primary outcome) and establish feasibility and acceptability, while also evaluating preliminary efficacy outcomes and EF change mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 7-12
* at least one caregiver/legal guardian able to participate (more permitted)
* experienced at least one episode of SITBs within the last month
* ability to attend weekly sessions in-person or via telehealth
* ability to attend baseline and 12-week assessments in-person.
* estimated verbal IQ of 70 or greater

Exclusion Criteria

* symptoms interfering with ability to participate in assessments/therapy (i.e., psychosis)
* estimated verbal IQ<70 or previous diagnosis of intellectual development disorder
* requiring inpatient psychiatric stabilization or high-intensity intervention to prevent hospitalization
* active substance use
* ward of the state

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Treatment Engagement | From enrollment to post-treatment at 12 weeks
  Number of treatment sessions completed at post-treatment
Feasibility of Retention | From enrollment to the end of treatment at 12 weeks
  % participants completing treatment (benchmark =≥ 80% participants considered treatment completers)
Feasibility of recruitment | Calculated at enrollment
  % recruitment targets met (benchmark = 52 preadolescents randomized to receive treatment)
Feasibility of Measurement | From enrollment to follow-up at 24 weeks
  % participants at each timepoint completing measures (target = ≥ 80% at each timepoint).
Perceived acceptability of intervention | From enrollment to the end of treatment at 12 weeks
  The Acceptability of Intervention Measure (AIM; Weiner et al., 2017) will be completed by preadolescents, caregivers, and therapists. The AIM is a 4-item measure assessing the extent to which stakeholders believe an intervention to be acceptable. Items are rated from 1 ("completely disagree") to 5 ("completely agree"), with higher scores indicating greater acceptability. The acceptability benchmark for all reporters is set at a mean score of 4 or greater.
Perceived Feasibility of Intervention | From enrollment to the end of treatment at 12 weeks
  The Feasibility of Intervention Measure (FIM; Weiner et al., 2017) will be completed by preadolescents, caregivers, and therapists. The FIM is a 4-item measures assessing the extent to which stakeholders believe an intervention to be feasible. Items are rated from 1 ("completely disagree") to 5 ("completely agree"), with higher scores indicating greater feasibility. The feasibility benchmark for all reporters is set at a mean score of 4 or greater.
Perceived Appropriateness of Intervention | From enrollment to the end of treatment at 12 weeks
  The Intervention Appropriateness Measure (IAM; Weiner et al., 2017) will be completed by preadolescents, caregivers, and therapists. The IAM is a 4-item measure assessing the extent to which stakeholders believe an intervention or to be appropriate. Items are rated from 1 ("completely disagree") to 5 ("completely agree"), with higher scores indicating greater appropriateness. The appropriateness benchmark for all reporters is set at a mean score of 4 or greater.

SECONDARY OUTCOMES:
Suicidal Ideation Intensity | From enrollment to 3-month follow-up at 24 weeks
  Measured using the Columbia Suicide and Self Injury Severity Rating Scale (C-SSRS; Posner et al., 2011), a brief interview that consists of sections that assess: suicidal ideation, ideation intensity, and suicidal behavior. The C-SSRS has strong convergent validity, sensitivity to change, predictive and incremental validity, and good internal consistency.
Readmission/Admission Rates | From enrollment to 3-month follow-up at 24 weeks
  Readmission/admission rates to the psychiatric ED or inpatient psychiatric hospitalization will be evaluated via caregiver report on the Brief form of the Services Assessment for Children and Adolescents (SACA; Horwitz et al., 2001), which will be supplemented with chart review.
Non-Suicidal Self-Injury | From enrollment to 3-month follow-up at 24 weeks
  Measured using an adapted version of the Self-Injurious Thoughts and Behaviors Interview (SITBI)-Short Form, Thoughts of NSSI and NSSI subscales (Nock et al., 2007), which assesses history and characteristics of NSSI thoughts and behaviors. First instance of engagement in NSSI after beginning treatment will be the outcome of most interest, but other outcomes assessed by the interview (e.g., frequency of NSSI thoughts) may be examined as well if rates of NSSI are very low.

OTHER OUTCOMES:
Anxiety Symptoms | From enrollment to 3-month follow-up at 24 weeks
  We will measure anxiety using the Revised Child Anxiety and Depression Scale (RCADS)-Short Version (Ebesutani et al., 2012; 2017), which is a 25-item measure of depression and anxiety symptoms that includes both parent-and self-report measures. Both versions are rated on a 5-point Likert scale, with higher scores indicating greater frequency of anxiety symptoms. Anxiety items are summed to yield a raw score, which is then converted to a t-score. The measure has good psychometric properties and treatment sensitivity (Ebesutani et al., 2012; 2017).
Depression Symptoms | From enrollment to 3-month follow-up at 24 weeks
  We will measure depression using the Revised Child Anxiety and Depression Scale (RCADS)-Short Version (Ebesutani et al., 2012; 2017), which is a 25-item measure of depression and anxiety symptoms that includes both parent-and self-report measures. Both versions are rated on a 5-point Likert scale, with higher scores indicating greater frequency of depression symptoms. Depression items are summed to yield a total raw score, which is then converted to a t-score. The measure has good psychometric properties and treatment sensitivity (Ebesutani et al., 2012; 2017).
Disruptive Behavior Symptoms | From enrollment to 3-month follow-up at 24 weeks
  We will measure disruptive behaviors using the Disruptive Behavior Disorders Scale (DBRS)-Parent Version (Fosco et al., 2023), a 45-item rating scale used to assess symptoms of inattention, hyperactivity-impulsivity, and oppositional defiant behavior among school-aged children. Items are rated on a 4-point scale, with higher scores indicating greater severity of symptoms.
Emotion Dysregulation--Reactivity | From enrollment to 3-month follow-up at 24 weeks
  Measured using the Emotion Dysregulation Inventory-Reactivity Short Form (EDI-R; Mazefsky et al., 2018; 2021), which includes a 7-item, caregiver report measure of emotional reactivity. Items are rated on a 5-point Likert scale, with higher scores indicating greater emotional reactivity.
Emotion Dysregulation--Dysphoria | From enrollment to 3-month follow-up at 24 weeks
  Measured using the Emotion Dysregulation Inventory-Dysphoria Short Form (EDI-D; Mazefsky et al., 2018; 2021), which is a 6-item, caregiver report measure of dysphoria in youth. Items are rated on a 5-point Likert scale, with higher scores indicating greater dysphoria.
Caregiver Report of Preadolescent Executive Functioning | From enrollment to 3-month follow-up at 24 weeks
  The Brief Rating Inventory of Executive Function 2nd Edition (BRIEF 2) --Parent Form (Gioia et al., 2015) is 63-item questionnaire with eight clinical scales designed to assess everyday behaviors associated with seven domains of EF. These scales are combined to form two broader indices (Behavioral Regulation and Metacognition) and a Global Executive Composite score. Items are rated on a 4-point scale, and sum scores for each scale and index are converted to t-scores, with higher t-scores indicating greater difficulties with executive functioning. The measure has strong psychometric properties, discriminates between typically developing and clinical populations, and is sensitive to change.
Behavioral Assessment of Executive Functioning and Distress Tolerance | From enrollment through post-treatment at 12 weeks
  Executive Function Challenge Task (EFCT; Kenworthy et al., 2014, 2020) is a "hot" measure of EF that uses a standardized protocol to assess flexibility and planning during several activities with an examiner that change rules or modalities. The EFCT has precise behavioral markers to guide scoring on a three-point scale and yields flexibility and planning raw scores that range from 0 to 8. The EFCT has good psychometric properties and demonstrated moderate associations with parent-reported EF and treatment-specific sensitivity to change (Kenworth et al., 2014; 2020).
Task-Based Assessment of Executive Functioning | From enrollment to the end of treatment at 12 weeks
  NIH toolbox Dimensional Change Card Sort test (DCCS; Kavanaugh et al., 2020; Zelazo et al., 2013). is a standard, lab-based, computerized task for assessing cognitive flexibility, will be administered as a computerized measure of EF. The DCCS has been validated in youth, does not demonstrate practice effects, and has excellent convergent validity.

IPD SHARING:
Plan to Share IPD: Yes
IPD from the randomized controlled trial will be shared with the NIMH National Data Archive.
Supporting Information: Study Protocol, SAP, ICF